CLINICAL TRIAL: NCT07387107
Title: Decreasing Stress Via Virtual Reality and Binaural Beats in Non-Clinical Adults: A Randomized Controlled Study.
Brief Title: Decreasing Stress Via Virtual Reality and Binaural Beats in Non-Clinical Adults
Acronym: DESTUD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Heart and Brain Research Group, Germany (Other)
Responsible Party: Principal Investigator, Dr. rer. nat. Dipl.-Psych. Marius Butz, Principal Investigator, Heart and Brain Research Group, Germany
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 110/21-DESTUD; DESTRESS (NCT05036538) (Other: Heart and Brain Research Group, Germany)
Record Dates: First submitted 2026-01-28; First posted 2026-02-04 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Stress; Relaxation; Virtual Reality; Binaural Beats
Keywords: Virtual Reality; Binaural Beats; Heart Rate Variability; Stress Reduction; Relaxation Intervention; Non-Clinical Population; Electrodermal Activity
MeSH Terms: interventions — Acoustic Stimulation

STUDY DESIGN:
Intervention Model Description: This study uses a randomized factorial, multi-arm design to evaluate the main effects and interaction of two intervention components: virtual reality-based natural environments (VR) and binaural auditory stimulation (binaural beats). Participants are randomly assigned to one of five parallel groups: (1) VR with binaural beats, (2) VR without binaural beats, (3) natural soundscapes with binaural beats, (4) natural soundscapes without binaural beats, or (5) a control condition without any relaxation intervention.
Masking Description: This is an open-label study. Due to the nature of the interventions, participants and investigators are not blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- VR + Binaural Beats (Experimental): Participants receive a virtual reality-based natural environment combined with binaural auditory stimulation for approximately 30 minutes.
  Interventions: Behavioral: Virtual Reality-Based Natural Environment; Behavioral: Binaural Auditory Stimulation
- VR Only (Experimental): Participants receive a virtual reality-based natural environment without binaural auditory stimulation for approximately 30 minutes.
  Interventions: Behavioral: Virtual Reality-Based Natural Environment
- Audio + Binaural Beats (Experimental): Participants receive natural soundscapes combined with binaural auditory stimulation without exposure to virtual reality for approximately 30 minutes.
  Interventions: Behavioral: Binaural Auditory Stimulation
- Audio Only (Experimental): Participants receive natural soundscapes without binaural auditory stimulation and without virtual reality exposure for approximately 30 minutes.
  Interventions: Behavioral: Auditory Stimulation
- Control (Experimental): Participants complete standardized control activities without any relaxation intervention for approximately 30 minutes.
  Interventions: Behavioral: Control Condition (No Relaxation Intervention)

INTERVENTIONS:
Behavioral: Virtual Reality-Based Natural Environment — Participants are exposed to immersive virtual reality-based natural landscapes using a head-mounted display for approximately 30 minutes. The content consists of non-animated 360° natural environments
  Arms: VR + Binaural Beats; VR Only
Behavioral: Binaural Auditory Stimulation — Participants receive auditory stimulation via headphones consisting of natural soundscapes combined with binaural beats. The binaural beat frequency is gradually reduced from the alpha range (10 Hz) to the delta range (1 Hz) over approximately 30 minutes.
  Arms: Audio + Binaural Beats; VR + Binaural Beats
Behavioral: Control Condition (No Relaxation Intervention) — Participants complete standardized control tasks without exposure to any relaxation intervention.
  Arms: Control
Behavioral: Auditory Stimulation — Participants receive auditory stimulation via headphones consisting of natural soundscapes over approximately 30 minutes.
  Arms: Audio Only

SUMMARY:
This study is a non-clinical substudy conducted within the DESTRESS research program (NCT05036538), which investigates the effects of relaxation interventions on physiological and psychological parameters. While the main DESTRESS trial focuses on cardiac surgical patients, this additional study arm examines the same interventions in a non-clinical adult population under controlled conditions, independent of disease-, surgery-, or medication-related influences.

Participants are randomly assigned to one of several experimental conditions and take part in a single approximately 30-minute session. Depending on group allocation, the session may include exposure to natural soundscapes, natural soundscapes combined with binaural beats, virtual reality-based natural environments, virtual reality combined with binaural beats, or a control condition without a relaxation intervention.

The primary aim of the DESTUD-Study is to assess the feasibility and potential stress-reducing effects of these non-pharmacological relaxation approaches in a non-clinical setting and to support the interpretation of findings from the clinical DESTRESS trial. Physiological responses, including heart rate variability and electrodermal activity, as well as self-reported stress measures, are collected before, during and after the conditions.

DETAILED DESCRIPTION:
This study is conducted as a non-clinical substudy within the DESTRESS research program (Decreasing preoperative stress to prevent postoperative delirium and postoperative cognitive decline in cardiac surgical patients: A randomized controlled trial on relaxation interventions via virtual reality and binaural beats; NCT05036538). In contrast to the main clinical trial, which investigates cardiac surgical patients, this study focuses on non-clinical adult participants who are not undergoing medical or surgical treatment and are not enrolled as patients of the Kerckhoff-Clinic Bad Nauheim (Germany).

The purpose of this substudy is to examine the effects of relaxation interventions under controlled conditions, independent of disease-related, perioperative, or pharmacological confounding factors. The results are intended to provide a reference framework for interpreting and contextualizing findings from the clinical DESTRESS trial.

Participants are randomly assigned to one of five experimental conditions: (1) natural soundscapes, (2) natural soundscapes combined with binaural beats, (3) virtual reality-based natural environments, (4) virtual reality-based natural environments combined with binaural beats, or (5) a control condition without any relaxation intervention. Each participant completes a single session lasting approximately 30 minutes.

During the intervention or control condition, physiological parameters, including heart rate variability and electrodermal activity, are continuously recorded using non-invasive sensors. Neurocognition and subjective stress levels are assessed using standardized tests and self-report questionnaires administered before and after the session.

This study aims to evaluate the feasibility, acceptability, and preliminary efficacy of virtual reality- and audio-based relaxation interventions in a non-clinical population. The findings are expected to contribute to a better understanding of the mechanisms and generalizability of stress-reduction approaches and to inform the interpretation of outcomes in the overarching DESTRESS research program.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years or older
2. Ability to understand study procedures and provide written informed consent
3. Sufficient proficiency in the German language to complete questionnaires and follow study instructions
4. Willingness to participate in a single approximately 60-minute study session

Exclusion Criteria:

1. Current or history of neurological or psychiatric disorders that may interfere with data collection (e.g., dementia, major depressive disorder, stroke, epilepsy)
2. Severe visual or hearing impairments that would limit the use of virtual reality equipment or headphones
3. Known cardiac arrhythmias or use of cardiac pacemakers/implantable devices that may interfere with heart rate variability measurements
4. Current use of psychoactive or cardiovascular medications that may significantly affect autonomic nervous system function
5. History of severe motion sickness, vertigo, or adverse reactions to virtual reality

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Change in High-Frequency Power of Heart Rate Variability (HF-HRV) | Pre- and post-intervention within a single 30-minute study session
  High-frequency (HF) power of heart rate variability will be used as an index of parasympathetic activity. The primary outcome is defined as the pre- to post-intervention change in HF-HRV measured continuously during the intervention or control condition.

SECONDARY OUTCOMES:
Change in Heart Rate Variability Parameters (RMSSD, NN50, pNN50, HF, HF%) | Pre- and post-intervention within a single 30-minute study session
  Changes in time- and frequency-domain heart rate variability parameters, including RMSSD, NN50, pNN50, HF power, and HF percentage, will be assessed during the intervention or control condition.
Change in Self-Reported Stress (Visual Analog Scale) | Pre- and post-intervention within a single 30-minute study session
  Self-reported stress levels will be assessed using a visual analog scale (VAS). The outcome is defined as the pre- to post-intervention change in perceived stress within the intervention or control condition.
Change in State Anxiety (STAI-6) | Pre- and post-intervention within a single 30-minute study session
  State anxiety will be assessed using the short form of the State-Trait Anxiety Inventory (STAI-6). The outcome is defined as the pre- to post-intervention change in anxiety scores within the intervention or control condition.
Change in Cognitive Flexibility (SKT) | Pre- and post-intervention within a single 30-minute study session
  Cognitive flexibility will be assessed using the Syndrom-Kurztest (SKT-7). The outcome is defined as the pre- to post-intervention change in test performance within the intervention or control condition.
Change in Verbal Fluency (Regensburger Word Fluency Test, RWT) | Pre- and post-intervention within a single 30-minute study session
  Verbal fluency will be assessed using the Regensburger Wortflüssigkeitstest (RWT). The outcome is defined as the pre- to post-intervention change in test performance within the intervention or control condition.
Change in Attention and Processing Speed (Trail Making Test A and B) | Pre- and post-intervention within a single 30-minute study session
  Attention and processing speed will be assessed using the Trail Making Test parts A and B (TMT A/B). The outcome is defined as the pre- to post-intervention change in test performance within the intervention or control condition.

CONTACTS AND LOCATIONS:
Overall Officials: Marius Butz, PhD, M.Sc., Principal Investigator — Heart&Brain Research Group, Kerckhoff-Clinic, Bad Nauheim, Germany